CLINICAL TRIAL: NCT04775121
Title: Classical Monocyte Kinetics in Chronic Myelomonocytic Leukemia
Acronym: MONOLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A01882-53; 2018/2774 (Other: CSET number)
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Myelomonocytic Leukemia

STUDY DESIGN:
Intervention Model Description: Deuterium glucose ingestion on a 3-hour period to label rapidly proliferating cells, followed by sequential collection of sorted classical monocytes on a 30-day period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Oral administration of 20 g Deuterium Glucose on a 3-hour period followed by sequential blood sampling to sort monocytes on a 30-days period of time
  Interventions: Other: Deuterium Glucose
- Healthy volunteers (Experimental): Oral administration of 20 g Deuterium Glucose on a 3-hour period followed by sequential blood sampling to sort monocytes on a 30-days period of time
  Interventions: Other: Deuterium Glucose

INTERVENTIONS:
Other: Deuterium Glucose — Oral administration of 20 g Deuterium Glucose on a 3-hour

SUMMARY:
To measure the rate of bone marrow release and the lifespan of classical monocytes in the peripheral blood of patients with a chronic myelomonocytic leukemia

ELIGIBILITY:
Inclusion Criteria for patients with CMML:

* Adult aged 18 years or over
* CMML diagnosis according to the WHO 2016 criteria
* Untreated patient or patient who did not receive a cytoreductive drug such as Hydroxyurea or an Erythropoiesis Stimulating Agent (ESA), or a growth factor, or Eltrombopag within the last 2 months or patient who did not receive a hypomethylating drug (Azacytidine or Decitabine) within the last 3 months
* Affiliated to a social security system or beneficiary of the same
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Able to comprehend the Information Sheet and willing to give written informed consent prior to any protocol-specific procedures performed
* Willing to allow the Investigator to review data from the hospital medical records
* For women of child-bearing age only, willingness to practice continuous effective contraception during the study. Women of childbearing potential must have a negative urine β-HCG pregnancy test within 15 days prior to the first administration of deuterium-labeled glucose. Sexually active male patients must agree to use condoms during the study. Also, it is recommended their women of childbearing potential partner use an effective method of contraception during the same period

Exclusion Criteria for patients with CMML:

* Severe anemia (Hb < 10 g/dL)
* Severe thrombocytopenia (Platelets < 50 G/L)
* Transfusion dependency
* Active or recent infection or febrile illness (<1 month)
* Currently active inflammatory or autoimmune condition
* Current systemic steroid therapy or other immunomodulatory drugs
* Recent vaccination (< 1 month)
* Recent surgery (< 1 month)
* Active malignant disease
* Renal disease (serum creatinine> 300µmol/L)
* Hepatic disease (transaminase levels >3x ULN)
* Severe or unstable cardiovascular disease
* Pregnancy or breastfeeding
* Other current active medical condition which the Investigator considers a risk for entry in the study
* Simultaneous participation in another concurrent research study that conflicts e.g. if it also involves blood sampling
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Inclusion Criteria of age-matched healthy donors:

* Volunteers aged 55 years or over
* Able and willing to comply with all study requirements
* Able to comprehend the Information Sheet and willing to give written informed consent prior to any protocol-specific procedures performed
* For women of child-bearing age only, willingness to practice continuous effective contraception during the study. Women of childbearing potential must have a negative urine β-HCG pregnancy test within 15 days prior to the first administration of deuterium-labeled glucose. Sexually active male patients must agree to use condoms during the study. Also, it is recommended their women of childbearing potential partner use an effective method of contraception during the same period.

Exclusion Criteria of age-matched healthy donors:

* Current treatment for any type of disease
* Current active medical condition
* Recent vaccination (< 1 month)
* Recent surgery (< 1 month)
* Pregnancy or breastfeeding
* Simultaneous participation in another concurrent research study that conflicts e.g. if it also involves blood sampling
* Subject under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Bone marrow release | up to 30 days
  To measure bone marrow release in the peripheral blood of patients with a chronic myelomonocytic leukemia and age-matched healthy volunteers

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Gustave Roussy, Villejuif, Val De Marne
  - Hôpital Saint Louis, Paris

IPD SHARING:
Plan to Share IPD: Undecided